CLINICAL TRIAL: NCT01255397
Title: Proposed Research Protocol For Male Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Amir Weiss, HaEmek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MF-001
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Male Infertility
Keywords: male infertility; natural cycle IVF; in-vitro fertilization; intrauterine inseminatio
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Male Infertility Protocol (Experimental)
  Interventions: Procedure: Male Infertility Protocol

INTERVENTIONS:
Procedure: Male Infertility Protocol — 1. Healthy women with a regular cycle between 28 and 35 days. For the man, an abnormal sperm exam.
  2. Daily US examinations from day 8 of the menstrual cycle. Excluding weekends.
  3. When the leading follicle is 14 mm she will be given 100 units puregon and orgalutran,once daily until the leading follicle is at least 16 mm at which point she will be given ovitrelle at 21:00.
  4. 35 hours after Ovitrelle at 8:00 the husband will present a sperm sample for analysis. A pelvic US will be done to the wife.
     1. If the follicle has collapsed than IUI will be performed
     2. It the total motile sperm count is above 5 million sperm/ml then IUI will be done
     3. If the total motile sperm count is below 5 million and the follicle has not collapsed, proceed to oocyte aspiration and ICSI
  6) ICSI and embryo transfer performed on the same day. 7) Luteal support: Endometrin 100 mg twice a day following IUI\ET until 6 weeks gestation Protocol can be repeated for up to 3 cycles per couple.

SUMMARY:
The purpose of this experiment is to test the feasibility of a minimally interventionist protocol for young couples with male factor infertility, which addresses the cause of infertility for these couples which is the inability of the sperm to fertilize the egg.Ultrasound monitoring of natural follicular development utilizing rFSH, GnRH antagonist and rHCG only for the final maturation. Single follicle aspiration and IUI or IVF/ICSI based on sperm charcteristics on the day of fertilization. Fertilized eggs transfered to the uterus on the same day as the aspiration.

ELIGIBILITY:
Inclusion Criteria:

1. Couples with "pure" male factor infertility of six months or more, defined as not pregnant in spite of being desirous of pregnancy for at least six months with normal sexual activity and no birth control. Primary and Secondary infertility included.
2. Abnormality of any one of the sperm parameters according to WHO or Kruger for concentration, motility or morphology.
3. Women aged 18 to 30 with a BMI between 18 and 30
4. Women who testify that they are healthy with regular menstrual cycles between 25-35 days per cycle.

Exclusion Criteria:

1. Uterine fibroids or ovarian cysts or tumors or suspected hydrosalpinx on US on prior fertility workup. Paraovarian simple cysts, OK.
2. Prior PID, abdominal or pelvic surgery or abnormal HSG if done.
3. Known allergy to medications used in protocol
4. Diagnosed or suspected genetic or psychiatric disease in either patient.
5. Azoospermia
6. Female partner with a history of infertility with another partner
7. Elevated FSH (over 10 units/L) in female partner if done.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01